CLINICAL TRIAL: NCT01632982
Title: Providing Psychosocial Interventions to Substance Abusers Via Mobile Technology
Brief Title: Mobile Psychosocial Interventions for MMT Clients
Acronym: MobileMMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mobile631; R01DA029630 (NIH)
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Opioid Abuse; Substance Abuse
Keywords: opioid abuse; substance abuse; methadone maintenance treatment; mobile technology; technology-based intervention; behavioral intervention; psychosocial treatment
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- standard treatment (Other): the standard drug counseling offered to patients in methadone maintenance treatment at the study site
  Interventions: Behavioral: standard treatment
- Mobile Therapeutic System (MTS) (Experimental): The Mobile Therapeutic System (MTS) is a novel, interactive, mobile phone-delivered psychosocial intervention designed to promote skills acquisition and reduce drug use among adults in methadone maintenance treatment
  Interventions: Behavioral: standard treatment; Behavioral: MTS (Mobile Therapeutic System)
- mobile control (Active Comparator): a mobile phone-based application that directs participants to the NIDA website's home page
  Interventions: Behavioral: standard treatment; Behavioral: mobile control

INTERVENTIONS:
Behavioral: standard treatment — the standard drug counseling offered to patients at the study site's methadone maintenance program
Behavioral: MTS (Mobile Therapeutic System) — a novel, interactive, mobile phone-delivered psychosocial intervention designed to promote skills acquisition and reduce drug use among adults in methadone maintenance treatment
  Arms: Mobile Therapeutic System (MTS)
Behavioral: mobile control — a mobile phone-based application that directs participants to the NIDA website's homepage
  Arms: mobile control

SUMMARY:
This study will develop and evaluate the preliminary efficacy and cost-effectiveness of a mobile phone-delivered psychosocial intervention for opioid-dependent adults (N=219) in methadone maintenance treatment (MMT). A three-arm, randomized clinical trial will evaluate the relative efficacy of: (1) standard MMT; (2) standard MMT plus the mobile intervention; and (3) a mobile-based control condition on the primary outcomes of treatment retention and opioid use (assessed via urine toxicology). If results are promising, this novel therapeutic tool may have a tremendous impact on improving access to and effectiveness of substance abuse treatment in a variety of other populations (and could also be adapted for an array of other behavioral health applications), while significantly limiting costs.

DETAILED DESCRIPTION:
This study will develop and implement a mobile technology-delivered psychosocial intervention for opioid-dependent adults in methadone maintenance treatment (MMT). This novel therapeutic system promises to be cost-effective and to enable the provision of flexible, on-demand therapeutic support outside of the formal treatment setting. The specific aims of this investigation are as follows: Aim 1: The investigators will develop a novel, interactive, evidence-based psychosocial intervention delivered via mobile phones, designed to promote skills acquisition and reduce illicit drug use. Specifically, our Mobile Therapeutic System (MTS) will offer key elements of a psychosocial intervention for substance use disorders of known efficacy (the Community Reinforcement Approach). Participants will be provided with unlimited daily prompts to encourage use of the program and will be able to access the application at any time and as much as they choose, within their natural environments. Our iterative development process will include input from focus groups with clients in methadone treatment (n=24), input from experts in the field, and feedback testing of a beta-version of the mobile phone-based program with clients in methadone treatment (n=30). Aim 2: The investigators will evaluate the efficacy of this mobile tool with participants entering MMT during the first three months of their treatment (n=219). The investigators will evaluate the relative preliminary efficacy of (1) standard treatment, (2) standard treatment plus MTS and (3) a mobile-based control condition on the primary outcomes of retention and opioid use (via urine toxicology) and secondary outcomes of other substance use (via urine toxicology and self-report), readiness to change drug use behavior, coping skills, opioid craving, HIV risk behavior, and psychosocial functioning during the 3-month intervention phase. Durability of effects will be examined at 1 and 3 month follow-ups. Aim 3: The investigators will perform an economic analysis of MTS in community-based MMT. The investigators will estimate the incremental costs and the incremental cost-effectiveness ratio (ICER) of MTS relative to standard care and the mobile control group. The primary ICER will be the incremental costs per increased abstinence time (the clinical measure of effectiveness) and the secondary ICER will be incremental costs per increased quality adjusted life year (QALY) (the economic measure of effectiveness). Cost data will be vital to future translational projects to disseminate effective mobile interventions in community systems. If results are promising, this novel therapeutic tool may have a tremendous impact on improving access to and effectiveness of substance abuse treatment in a variety of other populations (and could also be adapted for an array of other behavioral health applications), while significantly limiting costs.

ELIGIBILITY:
Inclusion Criteria:

* client enrolled in the study site's methadone maintenance program
* within the first month of initiating methadone maintenance treatment
* 18 years of age or older
* sufficient English-language ability to participate in informed consent process, complete study assessments and understand the text in mobile phone- delivered interventions

Exclusion Criteria:

* entering treatment at the study site with the intention of receiving a methadone-assisted withdrawal only
* evidence of an active psychiatric disorder requiring immediate intervention (e.g., suicidality, psychosis)
* evidence of significant mental illness that may preclude participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-11 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
treatment retention | 6 months
  participants' retention in methadone maintenance treatment (MMT)
opioid use | 6 months
  participants' illicit use of opioids, as measured by urine toxicology and self-report (self-report data collected via the timeline follow-back calendar assessment [TLFB])

SECONDARY OUTCOMES:
other substance use | 6 months
  participants' use of alcohol and drugs, as measured by urine toxicology and self-report (self-report data collected via the timeline follow-back calendar assessment [TLFB])
coping skills | 6 months
  participants' coping skills as measured by the Coping Strategies Scale (CSS)
readiness to change drug use | 6 months
  participants' readiness to change drug use, as measured by the Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES)
heroin/opioid craving | 6 months
  participants' craving for heroin and/or other opioids, as measured by the Heroin/Opiate Craving Questionnaire (HCQ)
HIV risk behavior | 6 months
  participants' HIV risk behavior as measured by the High Risk-Taking Behavior Scale (HRBS)
psychiatric and psychosocial functioning | 6 months
  participants' level of psychiatric functioning (as assessed by the Brief Symptom Inventory [BSI]) and psychosocial functioning (as assessed by the Addiction Severity Index [ASI])

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Acosta, Ph.D., Principal Investigator — National Development and Research Institutes (NDRI); Lisa A. Marsch, Ph.D., Principal Investigator — Dartmouth College; Honoria Guarino, Ph.D., Study Director — National Development and Research Institutes (NDRI)
Locations (1):
- Bridge Plaza Treatment and Rehabilitation Clinic, Long Island City, New York, United States